CLINICAL TRIAL: NCT06212076
Title: A Phase I/II, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamic Characteristics and Initial Anti-tumor Activity of IPG1094 in Patients With Advanced Solid Tumors
Brief Title: Phase I/II Study of IPG1094 in Advanced Solid Tumors Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Immunophage Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPG1094-C002
Record Dates: First submitted 2023-12-25; First posted 2024-01-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 (200 mg BID) (Experimental): Starting at 200mg BID cohort, 3 subjects will be enrolled. After 3 subjects completed DLT evaluation, the Safety Monitoring Committee (SMC) will review all available safety and PK/PD data from all treated subjects (DLT evaluable and non-DLT evaluable subjects), taking into consideration the dose-assignment recommendation based on 3+3 decision rule , to make the recommendation on the conduct of the study including the dose level and dose schedule for subsequent subjects.
  Interventions: Drug: IPG1094
- Cohort 2 (250 mg BID) (Experimental): Starting at 250 mg BID cohort, 3 subjects will be enrolled. After 3 subjects completed DLT evaluation, the Safety Monitoring Committee (SMC) will review all available safety and PK/PD data from all treated subjects (DLT evaluable and non-DLT evaluable subjects), taking into consideration the dose-assignment recommendation based on 3+3 decision rule , to make the recommendation on the conduct of the study including the dose level and dose schedule for subsequent subjects.
  Interventions: Drug: IPG1094
- Cohort 3 (NSCLC) (Experimental): Phase B is an expansion study to evaluate the anti-tumor efficacy and safety of IPG1094 in patients with non small cell lung cancer (specific tumor types will depend on the results of Part A), with 12 subjects enrolled. A sparse sampling approach for PK with 3 to 4 time points on Day 1 and 3 to 4 time points on Day 28 of Cycle 1, and pre-dose on Day 1 of Cycle 2 and every other cycle thereafter (for example, C4D1, C6D1, C8D1) to allow for population PK and exposure-response (efficacy and safety endpoints) analyses.
  Interventions: Drug: IPG1094
- Cohort 4 (TNBC) (Experimental): Phase B is an expansion study to evaluate the anti-tumor efficacy and safety of IPG1094 in patients with triple-negative breast cancer (specific tumor types will depend on the results of Part A), with 12 subjects enrolled. A sparse sampling approach for PK with 3 to 4 time points on Day 1 and 3 to 4 time points on Day 28 of Cycle 1, and pre-dose on Day 1 of Cycle 2 and every other cycle thereafter (for example, C4D1, C6D1, C8D1) to allow for population PK and exposure-response (efficacy and safety endpoints) analyses.
  Interventions: Drug: IPG1094
- Cohort 5 (head and neck cancer) (Experimental): Phase B is an expansion study to evaluate the anti-tumor efficacy and safety of IPG1094 in patients with head and neck cancer (specific tumor types will depend on the results of Part A), with 12 subjects enrolled. A sparse sampling approach for PK with 3 to 4 time points on Day 1 and 3 to 4 time points on Day 28 of Cycle 1, and pre-dose on Day 1 of Cycle 2 and every other cycle thereafter (for example, C4D1, C6D1, C8D1) to allow for population PK and exposure-response (efficacy and safety endpoints) analyses.
  Interventions: Drug: IPG1094
- Cohort 6 (brain glioma) (Experimental): Phase B is an expansion study to evaluate the anti-tumor efficacy and safety of IPG1094 in patients with brain glioma (specific tumor types will depend on the results of Part A), with 12 subjects enrolled. A sparse sampling approach for PK with 3 to 4 time points on Day 1 and 3 to 4 time points on Day 28 of Cycle 1, and pre-dose on Day 1 of Cycle 2 and every other cycle thereafter (for example, C4D1, C6D1, C8D1) to allow for population PK and exposure-response (efficacy and safety endpoints) analyses.
  Interventions: Drug: IPG1094

INTERVENTIONS:
Drug: IPG1094 — IPG1094 Activity: An inhibitor of macrophage migration inhibitory factor (MIF) Dosage form: Tablet Strength: 50 mg and 100 mg

SUMMARY:
This is a phase 1, open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) characteristics and initial anti-tumor activity of IPG1094 in patients with advanced solid tumors. The study will be conducted in two parts: dose escalation phase (Part A) and expansion phase (Part B).

DETAILED DESCRIPTION:
Part A:

In this phase, dose escalation will start from 200 mg and the present 2 dose cohorts are 200 mg BID and 250 mg BID. Up to 12 subjects are expected to be enrolled in this part. In each cohort, all subjects will receive a single oral dose of IPG1094, followed by a 3-day single-dose PK study period. If no significant toxicity occurs, subjects will receive consecutive daily doses (QD, 28 days/cycle) until disease progression, death, unacceptable toxicity, or withdrawal of informed consent (whichever comes first). The DLT evaluation period includes the single-dose PK study period and the first cycle of treatment (within 31 days after the first dose). The remaining subjects within the same cohort will be dosed if no significant safety signals are identified in the first subject in 3 days.

Starting at 200 mg cohort, 3 subjects will be enrolled initially at each subsequent dose cohort in accordance with the 3+3 dose-escalation design. After 3 subjects in each cohort completed DLT evaluation, the Safety Monitoring Committee (SMC) will review all available safety and PK/PD data from all treated subjects (DLT evaluable and non-DLT evaluable subjects), taking into consideration the dose-assignment recommendation based on 3+3 decision rule (as described in the table below), to make the recommendation on the conduct of the study including the dose level and dose schedule for subsequent subjects.

Part B:

After all subjects in Part A completed DLT evaluations, the SMC will review all available safety, PK/PD and efficacy data from all treated subjects, to recommend 1 dose level for Part B. Phase B is an expansion study to evaluate the anti-tumor efficacy and safety of IPG1094 in patients with several types of solid tumors, including but not limited to small cell lung cancer, triple-negative breast cancer, head and neck cancer, and melanoma (specific tumor types will depend on the results of Part A), with 12 subjects in each cohort. A sparse sampling approach for PK with 3 to 4 time points on Day 1 and 3 to 4 time points on Day 28 of Cycle 1, and pre-dose on Day 1 of Cycle 2 and every other cycle thereafter (for example, C4D1, C6D1, C8D1) to allow for population PK and exposure-response (efficacy and safety endpoints) analyses.

Subjects will receive consecutive doses (at the recommended schedule, 28 days/cycle) until disease progression, death, unacceptable toxicity, or withdrawal of informed consent (whichever comes first).

The RP2D will be established by taking into consideration of the PK/PD profiles, safety and efficacy data from both Part A and Part B.

The anti-tumor activity will be evaluated according to the response evaluation criteria in solid tumors version 1.1 (RECIST v1.1). Efficacy assessments will be performed at the screening (within 28 days prior to first administration) and every 2 cycles (8 weeks±7 days) until disease progression, death, withdrawal of informed consent, or study discontinuation. Subjects who discontinue treatment for reasons other than disease progression or death should continue with imaging assessments per protocol-defined schedule until disease progression, death, starting new anti-tumor therapies or withdrawal of informed consent, whichever occurs first. Subjects may be contacted via phone for vital status every 3 months post the last dose until death, withdrawal of informed consent, loss to follow-up or study discontinuation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

1. Male or female aged ≥ 18 years.
2. In Part A:

   Subjects must have a histological diagnosis of locally advanced or metastatic malignant solid tumors, and that is not amenable to curative surgical and/or locoregional therapies;

   In Part B:

   Subjects must have a histological diagnosis of locally advanced or metastatic malignant solid tumors, and that is not amenable to curative surgical and/or locoregional therapies (tumor types in Part B will include but not limited to small cell lung cancer, triple-negative breast cancer, head and neck cancer, and melanoma).
3. Subjects must have failed or have been intolerant to established standard therapies, or standard therapies did not exist or were no longer effective for a given tumor type, or in the opinion of the investigator have been considered ineligible for a particular form of standard therapy on medical grounds.
4. Subjects must have at least one evaluable lesion according to RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
6. Life expectancy ≥ 12 weeks.
7. Subjects must have adequate organ and bone marrow function (no hematopoietic growth factor, blood transfusion, or platelet therapy within 2 weeks before the screening and during the screening):

   * Complete blood count (CBC): neutrophils ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 9.0 g/dL.
   * Liver function: total bilirubin ≤ 1.5 × ULN; ALT/AST ≤ 2.5 × ULN without liver metastasis; ALT/AST ≤ 5 × ULN with liver metastasis;
   * Coagulation: International normalized ratio (INR) ≤ 1.5 × ULN and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (for patients undergoing anticoagulant therapy. The investigator will judge that the INR and APTT are within a safe treatment range);
   * Renal function: creatinine clearance > 50 mL/min (calculated using the Cockcroft-Gault formula) in the condition of creatinine level > ULN; urine protein qualitative ≤ 1 + (if ≥ 2+, 24 hours of urine protein test is required, if 24 hours urine protein <1 g, then allowed to enroll);
   * Adequate cardiac function left ventricular ejection fraction (LVEF) > 50% for 2 dimensional cardiac ultrasound.
8. Women of childbearing potential (WOCBP) and fertile males with WOCBP partners must use highly effective contraception throughout the study (from first dose and through 28 days after final dose of study drug).
9. Subjects must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent form that under regulatory and institutional guidelines, and this must be obtained before the performance of any protocol-related procedures.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Subjects who received anti-tumor therapy (except for mitomycin, nitrosourea, and fluorouracil oral drugs) within 4 weeks before the first dose, including but not limited to chemotherapy, radiotherapy (palliative radiotherapy is completed at least 2 weeks before the first dose can be enrolled), targeted therapy or immunotherapy.

   Note: Mitomycin and nitrosourea have been treated within 6 weeks after the last dose; oral fluorouracil such as tegafur and capecitabine has been treated within 2 weeks after the last dose.
2. Subjects who have previous toxicity of anti-tumor therapy that has not been returned to level 0 or 1. (Alopecia, chemotherapy-induced peripheral neurotoxicity and ototoxicity ≤ Grade 2 can be enrolled).
3. Subjects who received CYP3A4 strong inhibitors or CYP3A4 strong inducers (see https://drug-interactions.medicine.iu.edu/MainTable.aspx) within 14 days prior to the first dose and the subjects who need to continue using these drugs throughout the study.
4. Subjects who received clinical intervention for biliary obstruction 14 days prior to the first dose or the investigator judges that the symptoms had not resolved or required anti-infective treatment.
5. Subjects who had clinically uncontrollable pleural effusion, ascites, or pericardial effusion within 2 weeks prior to the first dose.
6. Subjects who have symptomatic brain metastases or spinal cord compression. Subjects who have previously treated for brain metastases, if the clinical condition is stable and imaging evidence does not show disease progression within 4 weeks prior to the first dose and do not need corticosteroid treatment within 2 weeks prior to the first dose, can be enrolled.
7. Subjects who have active bacterial or fungal infections (≥ Grade 2) that required systemic treatment within 14 days prior to the first dose.
8. Subjects who participated in any other study in which receipt of an investigational new drug, or investigational device occurred within 28 days or 5 half-lives (whichever is shorter) of the first dose of the study drug.
9. Receiving systemic steroid therapy (> 10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study drug.
10. Subjects who have a chronic or active infection requiring systemic therapy.
11. Subjects who have gastrointestinal disorders that will affect oral administration or the investigator judges that the absorption of IPG1094 will be interfered.
12. Known or suspected allergy or hypersensitivity to any component of IPG1094.
13. Subjects who received a diagnosis of, and/or tested positive at screening for human immunodeficiency virus (HIV).
14. Subjects with positive Hepatitis B surface antigen [HBsAg] test, except for subjects who have negative HBsAg test and positive Hepatitis B core antibody [HBcAb] test combined with negative HBV DNA test at screening.
15. Co-infection of hepatitis B virus (HBV) and hepatitis C virus (HCV), subjects with a history of HCV infection but who are negative for HCV RNA by PCR will be considered non-infected with HCV.
16. Active other malignancy requiring treatment with the exception of any of the following:

    * Adequately treated basal cell carcinoma;
    * Squamous cell carcinoma of the skin, or in situ cervical cancer;
    * Low-risk prostate cancer (i.e. Gleason score < 7 and prostate specific antigen < 10 ng/mL); or
    * Any other cancer from which the individual has been disease-free for ≥ 5 years.
17. Subjects who have clinically significant cardiovascular diseases that occurred 6 months prior to enrollment. Cardiovascular diseases include, but not limited to follows:

    * Acute myocardial infarction;
    * Severe/unstable angina;
    * Cerebrovascular accident or transient ischemic attack;
    * Congestive heart failure (New York Heart Association > Class II);
    * Arrhythmias that require antiarrhythmic treatment except for beta blockers or digoxin;
    * Repeated ECG with QTc interval ≥ 470 msec regardless of sex (corrected according to Fridericia's formula);
    * High blood pressure that cannot be controlled by antihypertensive drugs (systolic blood pressure > 150 mm Hg, diastolic blood pressure > 100 mmHg).
18. Subjects who are receiving warfarin (low-dose warfarin as 2 mg/day is acceptable); or receiving antiplatelet anticoagulant therapy (aspirin at dose ≥300 mg/day, clopidogrel at dose ≥75 mg/day).
19. Major surgery or significant traumatic injury occurring within 28 days prior to the first dose of the study drug. If major surgery occurred > 28 days prior to the first dose of the study drug, the individual must have recovered adequately from the toxicity and/or complications from the intervention prior to the first dose of the study drug.
20. Female subjects in pregnancy or lactation.
21. Having difficulty in venous blood collection. Any other circumstances, in the opinion of the investigator, that may affect the subject's informed consent or adherence to the protocol, or that the subject's participation in the study may affect the outcome of the study or their own safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2027-07-09 (Estimated); Study Completion 2027-07-09 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | Up to 6 months
  Safety (AE occured over grade 3 in Subjects)
Primary endpoint | Up to 2 months
  Tolerability (AE occured over grade 3 in Subjects)
Primary endpoint | Up to 3 months
  maximum tolerated dose (MTD)
Primary endpoint | Up to 8 months
  recommended phase 2 dose (RP2D)

SECONDARY OUTCOMES:
Secondary endpoint 1 | Up to 6-8 months
  Pharmacokinetic of IPG1094: Maximum Plasma Concentration [Cmax], etc,
Secondary endpoint 2 | Up to 6-8 months
  Anti-tumor activity of IPG1094: RECIST 1.1 evaluation

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai GoBroad Cancer Hospital China Pharmaceutical University, Shanghai

IPD SHARING:
Plan to Share IPD: No